CLINICAL TRIAL: NCT05470933
Title: A Phase Ⅰ Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Antitumor Activity of WJ01075 Tablets in Oral Dose Escalation and Expansion in Patients With Advanced Solid Tumors
Brief Title: A Study Explore WJ01075 Tablets in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminate the study and close the research center based on strategic changes in product development, unrelated to drug safety.
Sponsor: Suzhou Junjing BioSciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS124-001-I
Record Dates: First submitted 2022-07-07; First posted 2022-07-22 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: Single Group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WJ01075 tablets (Experimental): Once a week (QW).
  Interventions: Drug: WJ01075

INTERVENTIONS:
Drug: WJ01075 — Phase Ia: Dose Escalation Accelerated titration (the first two dose groups) and "3 + 3" combination (the subsequent dose group) were used for dose escalation.
  Phase Ib: Dose Expansion and Cohort Expansion The actual dose, dosing schedule (including combination) and indication selection will be evaluated based on the results of existing trials.

SUMMARY:
This is a phase I study to Investigate the safety and tolerability, DLT(Dose limited toxicity), MTD(Maximum tolerated dose), and RP2D(Recommended phase II dose) of WJ01075 tablets in patients with advanced malignant solid tumors, including phase Ia (dose escalation phase) and Phase Ib (dose expansion phase,cohort expansion phase).The study includes screening, treatment and follow-up periods.

In phase Ia, accelerated titration (the first two dose groups) and "3 + 3" combination (the subsequent dose group) were used for dose escalation.

In phase Ib, specific dose groups will be selected for dose expansion according to PK(Pharmacokinetics) and safety data of different dose groups in dose escalation phase.It is planned that SMC(Safety Monitoring Committee) will select one or more dose groups based on previous data for cohort expansion studies to further determine RP2D, safety tolerability and initial efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with advanced malignant solid tumors clearly diagnosed pathologically and/or cytologically, who have failed to receive standard treatment, or who currently do not/or refuse standard treatment, or who are intolerant to standard treatment;
2. Patient must have at least one measurable lesion as defined per RECIST v1.1;
3. Aged between 18 and 75 (including 18 and 75), male and female patients;
4. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score ≤1;
5. Life expectancy ≥ 3 months;
6. The functions of patients' major organs were basically normal, and the laboratory tests performed within 7 days prior to the first administration of study drugmet the following criteria, Patients must not have required a blood transfusion or growth factor support within 14 days before the examination:

   Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤2.5 × Upper limit of Normal (ULN); Total Bilirubin≤ 1.5×ULN; International Normalized Ratio (INR) ≤1.5; Creatinine ≤ 1.5 × ULN, and Creatinine Clearance Rate (calculated by Cockcroft-Gault formula) ≥ 50 mL/min; Hemoglobin (Hg) ≥ 90g/L; Platelets ≥ 100×10⋀9/L; Absolute Neutrophil Count(ANC) ≥ 1.5×10⋀9/L
7. Fertile women must confirm a negative blood pregnancy test within 7 days prior to the first administration of study drug;All enrolled patients (both male and female) are required to use adequate and effective contraceptive measures throughout the treatment period and within 3 months after the end of treatment;
8. Those who voluntarily participate in the study and sign the written Informed Consent Form upon full informed consent.

Exclusion Criteria:

1. Prior treatment with XPO1 inhibitors;
2. Have a history of allergy to any component or excipient of WJ010175 tablets;
3. Patient with a primary malignancy other than the tumor treated in the study within 5 years prior to the first administration of study drug (exceptions include cured malignancies that did not recur within 3 years prior to enrollment;Basal cell and squamous cell carcinoma completely resected;Complete excision of any type of carcinoma in situ, etc.);
4. Received other anti-tumor therapies, including but not limited to chemotherapy, radiotherapy, targeted therapy, immunotherapy and other anti-tumor therapies (such as anti-tumor traditional Chinese medicine), within 4 weeks or 5 half-life periods (whichever is longer) prior to the first administration of study drug;Or long-term treatment with potent CYP1A2 inhibitors, potent CYP3A4 inducers and potent CYP3A4 inhibition;
5. Thrombosis or embolism occurred within 6 months prior to the first administration of study drug;
6. Received medium or major surgical treatment within 4 weeks prior to the first administration of study drug, other than diagnostic biopsy ;
7. Any of the following conditions within 6 months prior to the first administration of study drug: New York Cardiology Association (NYHA) > Grade II cardiac insufficiency, congestive heart failure, severe/unstable angina pectoris (symptoms of resting angina pectoris), myocardial infarction, arrhythmias requiring treatment, uncontrolled hypertension or hypertensive crisis or hypertensive encephalopathy;
8. Adverse events and/or complications caused by previous treatment are not relieved to < Level 2 (per NCI-CTCAE V5.0);Any level of hair loss/pigmentation and long-term toxicity caused by other treatment, other than those that the investigator diagnosiss cannot be recovered and do not affect study administration or compliance and patient safety;
9. Patient with central nervous system metastasis or tumors originating in the central nervous system;,
10. Patient with grade ≥ 2 neuropathy (per NCI-CTCAE V5.0);
11. Severe infections requiring antibiotic treatment within 14 days prior to the first administration of study drug ( > CTCAE Grade 2 ), such as severe pneumonia, bacteremia, infection complications requiring hospitalization;
12. Uncontrolled pericardial effusion, pleural effusion or clinically obvious moderate to severe abdominal effusion during screening is defined as meeting the following criteria: having clinical symptoms and detectable thoracic and abdominal effusion during physical examination;Or in the screening process, the thoracoabdominal effusion needs to be punctured pumping liquid and/or intravenously administered;
13. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
14. Patient has serious psychological or mental abnormalities affecting the compliance of the subjects to participate in the study;
15. With active Hepatitis B, or Hepatitis C, or Human Immunodeficiency Virus positive [HIV (+)] and syphilis antibody (+);Note: Hepatitis B virus surface Antigen (HBsAg) or core antibody (HBcAb) positive should be tested for HBV-DNA, and HBV-DNA should be below the lower limit of the reference range.Patients who are positive for Hepatitis C virus Antibody (HCV Ab) will be tested for HCV RNA and can be enrolled if they are below the upper limit of normal.
16. With Gastrointestinal dysfunction that may affect drug absorption (e.g., intestinal obstruction, inability to swallow tablets, malabsorption syndrome, uncontrollable nausea or vomiting, etc.);
17. Pregnant or lactating women or men who still have reproductive needs;
18. Other conditions that the investigator considers to be ineligible for inclusion, including but not limited to subjects whose body weight is less than ideal and who are expected to be significantly affected by weight change as determined by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Dose limited toxicity (DLT) | 3 years
  incidence and severity of Dose limited toxicity(DLT);
Adverse event (AE) | 3 years
  incidence and severity of adverse event (AE), Abnormal changes in laboratory and other tests of clinical significance;
Serious adverse event (SAE) | 3 years
  incidence and severity of Serious adverse event (SAE);
Maximum tolerated dose (MTD) | 2 years
  Maximum tolerated dose (MTD)
Recommended phase II dose (RP2D) | 2 years
  Recommended phase II dose (RP2D)

SECONDARY OUTCOMES:
Objective response rate(ORR) | 2 years
  Efficacy endpoints: Objective response rate(ORR) per RECIST v1.1
Duration of response (DOR) | 2 years
  Efficacy endpoints: Duration of response (DOR) per RECIST v1.1
Disease control rate (DCR) | 2 years
  Efficacy endpoints: Disease control rate (DCR) per RECIST v1.1
Time to response(TTR) | 2 years
  Efficacy endpoints: Time to response(TTR) per RECIST v1.1
Progression-free survival (PFS) | 2 years
  Efficacy endpoints: Progression-free survival (PFS) per RECIST v1.1
Overall survival (OS) | 2 years
  Efficacy endpoints: Overall survival (OS) per RECIST v1.1
Peak time(Tmax) | 2 years
  Pharmacokinetic (PK) parameter : Peak time(Tmax) after a single dose;
Maximum plasma concentration (Cmax) | 2 years
  Pharmacokinetic (PK) parameter : Maximum plasma concentration (Cmax) after a single dose;
Clearance rate (CL/F) | 2 years
  Pharmacokinetic (PK) parameter : Clearance rate (CL/F) after a single dose;
Apparent volume of distribution (Vd/F) | 2 years
  Pharmacokinetic (PK) parameter : Apparent volume of distribution (Vd/F) after a single dose;
Area under blood concentration - time curve (AUC) | 2 years
  Pharmacokinetic (PK) parameter : Area under blood concentration - time curve (AUC) after a single dose;
Elimination rate constant (λz) | 2 years
  Pharmacokinetic (PK) parameter : Elimination rate constant (λz) after a single dose;
Elimination half-life time ( t1/2) and other parameters | 2 years
  Pharmacokinetic (PK) parameter : Elimination half-life time ( t1/2) and other parameters after a single dose;
Steady state valley concentration(Cssmin) | 2 years
  Pharmacokinetic (PK) parameter : Steady state valley concentration(Cssmin) after repeated administration;
Steady state peak concentration(Cssmax) | 2 years
  Pharmacokinetic (PK) parameter : Steady state peak concentration(Cssmax) after repeated administration;
Average steady-state plasma concentration(Css-av) | 2 years
  Pharmacokinetic (PK) parameter : Average steady-state plasma concentration(Css-av) after repeated administration;
Elimination half-life time ( t1/2) | 2 years
  Pharmacokinetic (PK) parameter : Elimination half-life time ( t1/2) after repeated administration;
Steady state Area under blood concentration - time curve(AUCss) | 2 years
  Pharmacokinetic (PK) parameter : Steady state Area under blood concentration - time curve(AUCss) after repeated administration;
Fluctuation coefficient (DF) | 2 years
  Pharmacokinetic (PK) parameter : Fluctuation coefficient (DF) after repeated administration;
Steady-state distribution volume(Vss ) | 2 years
  Pharmacokinetic (PK) parameter : Steady-state distribution volume(Vss ) after repeated administration;
Accumulation coefficient (AR) and other parameters | 2 years
  Pharmacokinetic (PK) parameter : Accumulation coefficient (AR) and other parameters after repeated administration;

CONTACTS AND LOCATIONS:
Locations (1):
- Harbin Medical University Cancer Hospital, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No